CLINICAL TRIAL: NCT01021878
Title: A Study to Evaluate the Effects of Icodextrin vs 2.5% Dianeal Used for the Long Dwell in Apd: a Randomized, Open-label Clinical Trial to Analyse the Insulin Resistance Using the Homa Index in Prevalent, Non-diabetic Patients
Brief Title: Study to Evaluate the Effects Icodextrin Versus Dianeal on Insulin Resistance in Nondiabetic Automated Peritoneal Dialysis Patients
Acronym: STARCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontifícia Universidade Católica do Paraná (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Roberto Pecoits-Filho, MD, PhD, FASN, Pontifícia Universidade Católica do Paraná
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUCPR 01
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Disorders Associated With Peritoneal Dialysis
Keywords: Peritoneal dialysis; Renal replacement therapy; Dialysis solutions; Icodextrin
MeSH Terms: interventions — Icodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- icodextrin (Experimental): glucose sparing alternative dialysis solution
  Interventions: Other: icodextrin
- dextrose (Active Comparator): dianeal, Control group, standard treatment
  Interventions: Other: Dianeal

INTERVENTIONS:
Other: icodextrin — glucose sparing dialysis solution
  Other Names: Extraneal
  Arms: icodextrin
Other: Dianeal — glucose based dialysis solution
  Arms: dextrose

SUMMARY:
1. LOCATION OF STUDY: Multicentric study in Brazil.
2. PURPOSE OF THE STUDY: To measure changes in HOMA index when non-diabetic patients in APD were exposed to 7,5% Icodextrin for the long-dwell; and to compare such changes with those produced by 2,5% glucose for the long-dwell.
3. PRIMARY OUTCOME: The primary efficacy outcome was to measure HOMA index to set the differences with regard to baseline values of this variable for the two groups as well as in each group, which showed control of the glucose metabolism.

STAGE OF THE STUDY : Phase IV postmarket study

DESIGN: Randomized, open-label, multicenter study. Patients were randomized to receive either to Extraneal (7,5% Icodextrin) or 2.5% Dianeal during the long-dwell.

SAMPLE SIZE: Randomization Upon completion of the study TOTAL: 120 60 ExtranealTM 60 30 Dianeal® 60 30

Duration: 1 year.

DETAILED DESCRIPTION:
1. SUMMARY OF THE STUDY

1.1 PROTOCOLE TITLE : A RANDOMIZED, OPEN-LABEL CLINICAL TRIAL TO EVALUATE THE EFFECTS OF ICODEXTRIN Vs 2,5% DIANEAL USED FOR THE LONG-DWELL ON HOMA INDEX IN PREVALENT, NON-DIABETIC, PATIENTS IN AUTOMATED PERITONEAL DIALYSIS (APD)

1.2 MAIN RESEARCHERS: Roberto Pecoits Filho, Thyago P. Moraes

1.3 LOCATION OF STUDY: Multicentric study in Brazil.

1.4 PURPOSE OF THE STUDY: To measure changes in HOMA index when non-diabetic patients in APD were exposed to 7,5% Icodextrin for the long-dwell; and to compare such changes with those produced by 2,5% glucose for the long-dwell.

1.5 PRIMARY OUTCOME: The primary efficacy outcome was to measure HOMA index to set the differences with regard to baseline values of this variable for the two groups as well as in each group, which showed control of the glucose metabolism.

1.6 SECONDARY OUTCOMES:

1.6.1 Other efficacy outcomes were total UF, long-dwell UF, and preprandial glycemia (taken first in the morning before breakfast), serum insulin levels and glycated haemoglobin.

1.6.2 The incidence of adverse events will be measured as a safety outcome.

1.7 STAGE OF THE STUDY : Phase IV postmarket study

1.8 DESIGN: Randomized, open-label, multicenter study. Patients were randomized to receive either to Extraneal (7,5% Icodextrin) or 2.5% Dianeal during the long-dwell.

1.9 SAMPLE SIZE: Randomization Upon completion of the study TOTAL: 100 60 ExtranealTM 50 30 Dianeal® 50 30

1.12 PHARMACEUTICAL FORM, ROUTE OF DE ADMINISTRATION AND DOSAGE

ExtranealTM (7.5% Icodextrin) solution for Peritoneal Dialysis:

It is labelled as "solution for dialysis" to be administered within the study for a period of one (1) year.

Available in 2 liter bags of peritoneal dialysis solution (Twin Bag) for CAPD, this product will be used during the long-dwell.

Dianeal® PD4 (2.5% Dextrose) solution for Peritoneal Dialysis:

It is labelled as 2.27% glucose-based "solution for dialysis", to be administered within the study for a period of one (1) year.

Available in 2 and 2.5 liter bags of peritoneal dialysis solution (Twin Bag) for CAPD, this product will be used during the long-dwell.

Duration: 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 1.10.1 Older than 18 years old.
* High PET value, average-high or average-low.
* Cause of renal chronic disease other than diabetes mellitus.
* Patient in APD
* Prevalent patient in APD (defined as at least 90 total days of dialysis therapy)

Exclusion Criteria:

* Not willing to participate.
* A Charlson comorbidity index >7, or a life expectancy < 12 months as assessed by the treating physician.
* Positive VIH.
* Episodes of peritonitis during the month preceding the randomization.
* Significant cardiovascular, metabolic or infectious complications during the month preceding the randomization.
* Patients with active cancer.
* Patients with known allergies to corn starch polymers.
* Patients who are unable to provide an informed consent because of significant psychiatric disorder or mental illness
* Patients not meeting adequacy goals several months after the change in the dosage regime.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pecoits-Filho, MD, PhD, Principal Investigator — Pontificia Universidade Catolica do Parana
Locations (8):
- Brazil (8):
  - Hospital São João de Deus, Divinópolis, Minas Gerais
  - Universidade Federal de Uberlândia, Uberlândia, Minas Gerais
  - Clinica de Doencas Renais, Curitiba, Paraná
  - Instituto do Rim de Curitiba, Curitiba, Paraná
  - Nefroclinica de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Clinese, Aracaju, Sergipe
  - Universidade Estadual Paulista, Botucatu, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo, São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Icodextrin: glucose sparing alternative dialysis solution
  icodextrin: glucose sparing dialysis solution
  N=33
- Dextrose: Control group, standard treatment
  Dianeal: glucose based dialysis solution
  N=27
Period: Overall Study
Arm/Group | Icodextrin | Dextrose
Started | 33 | 27
Completed Follow-up | 17 | 17
Completed | 17 | 17
Not Completed | 16 | 10
Not completed — Lost to Follow-up | 4 | 3
Not completed — Death | 0 | 1
Not completed — Adverse Event | 6 | 5
Not completed — Transplantation | 6 | 1

BASELINE CHARACTERISTICS:
Population: From October 2009 to February 2012 60 patients were randomly assigned to the intervention (n=33) or the control (n=27) group. Completed follow-up was achieved for 34 patients, of which 17 of the control and 17 of the study group.
Groups:
- Dextrose: Control group, standard treatment
  Dianeal: glucose based dialysis solution
- Total: Total of all reporting groups
Arm/Group | Icodextrin | Dextrose | Total
Number analyzed (Participants) | 33 | 27 | 60
Age, Continuous [Median (Standard Deviation); unit: years] | 50.1 (15.5) | 54.1 (17.4) | 52.1 (16.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 15 | 12 | 27
Region of Enrollment [Number; unit: participants]
  Brazil | 33 | 27 | 60
HOMA index [Mean (Standard Deviation); unit: IR score] | 2.10 (1.10) | 1.77 (1.00) | 1.95 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted HOMA Index Score at 3 Months Using Baseline Values as a Covariate and Groups as the Fixed Factor
Description: Adjusted HOMA index score at 3 months using baseline values as a covariate and groups as the fixed factor. HOMA index was calculated as follows:
  (fasting glucose(mg/dl) x fasting serum insulin (μU/mL))/405
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: IR score
Arm/Group | Icodextrin | Dextrose
Number analyzed (Participants) | 33 | 27
IR score | 1.49 [1.23 to 1.74] | 1.89 [1.62 to 2.17]

2. Secondary Outcome: Oral Fasting Serum Glucose
Description: Serum glucose measured in oral fasting but not peritoneal fasting.
  For this outcome we compared groups using analysis of covariance (ANCOVA) using the baseline values as covariate, groups as the fixed factor and the value obtained at 90 days as the dependent variable. Significance level for alpha was setting at < 0.05.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Icodextrin | Dextrose
Number analyzed (Participants) | 33 | 27
mg/dl | 92.8 (20.0) [87.5 to 98.2] | 94.5 (17.9) [88.7 to 100.2]

3. Secondary Outcome: Serum Insulin
Description: Serum insulin was log-transformed to meet all criteria for ANCOVA. The baseline value was treated as covariate, groups as the fixed factor and the serum insulin at 3 months as the dependent variable. Serum insulin was measured in oral fasting by chemioluminescense.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: log(mmol/L)
Groups:
- Icodextrin: glucose sparing alternative dialysis solution
  icodextrin: glucose sparing dialysis solution
  There were a total of 25 adverse events reported of which 10 in the control group and 15 in the intervention group. Six were considered a severe event, 4 in the control group and 2 in the intervention group.
- Dextrose: Control group, standard treatment
  Dianeal: glucose based dialysis solution
  There were a total of 25 adverse events reported of which 10 in the control group and 15 in the intervention group. Six were considered a severe event, 4 in the control group and 2 in the intervention group.
Arm/Group | Icodextrin | Dextrose
Number analyzed (Participants) | 33 | 27
log(mmol/L) | 0.79 [0.70 to 0.87] | 0.90 [0.81 to 0.98]

4. Secondary Outcome: Glycated Hemoglobin
Description: Adjusted glycated hemoglobin was obtained and compared between groups using analysis of covariance (ANCOVA). The baseline values of HbA1c was used as covariate, the groups as the fixed factor and the value obtained at 90 days as the dependent variable.
  Glycated hemoglobin was measured by high-performance liquid chromatography.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: percentage of haemoglobin
Arm/Group | Icodextrin | Dextrose
Number analyzed (Participants) | 33 | 27
percentage of haemoglobin | 4.97 [4.73 to 5.21] | 4.86 [4.62 to 5.10]

5. Secondary Outcome: Total Ultrafiltration
Description: Total ultrafiltration obtained in 24 hours was obtained and compared between groups using analysis of covariance (ANCOVA). The baseline values of total ultrafiltration was used as covariate, the groups as the fixed factor and the value obtained at 90 days as the dependent variable.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: millilitre
Arm/Group | Icodextrin | Dextrose
Number analyzed (Participants) | 33 | 27
millilitre | 958 [818 to 1097] | 656 [517 to 795]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Patients were trained to report adverse effects immediately. Otherwise, adverse effects were checked every other week.
Arm/Group | Icodextrin | Dextrose
Serious Adverse Events (participants affected / at risk) | 4/33 | 5/27
Other Adverse Events (participants affected / at risk) | 1/33 | 1/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Icodextrin (N=33) | Dextrose (N=27)
Death (Infections and infestations) | 0 | 1 — Sepsis
Peritonitis (Infections and infestations) | 2 | 2 — Peritonitis related to Peritoneal dialysis
Exit-site infection (Skin and subcutaneous tissue disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Icodextrin (N=33) | Dextrose (N=27)
Ultrafiltration Failure (General disorders) | 0 | 1
Hernia (Musculoskeletal and connective tissue disorders) | 1 | 0
gastroesophageal reflux (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No